CLINICAL TRIAL: NCT05577195
Title: UNLOAD ECMO - Left Ventricular Unloading to Improve Outcome in Cardiogenic Shock Patients on VA-ECMO - a Prospective, Randomized, Controlled, Multi-center Trial
Brief Title: Left Ventricular Unloading to Improve Outcome in Cardiogenic Shock Patients on VA-ECMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNLOAD ECMO
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Cardiogenic Shock
Keywords: Active left ventricular unloading; VA-ECMO; Impella; Cardiogenic shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impella + VA-ECMO (Experimental)
  Interventions: Device: Impella; Device: VA-ECMO
- VA-ECMO only (Active Comparator)
  Interventions: Device: VA-ECMO

INTERVENTIONS:
Device: Impella — To provide active left ventricular unloading in the experimental arm
  Arms: Impella + VA-ECMO
Device: VA-ECMO — To provide circulatory support in both arms

SUMMARY:
Prospective, multi-center, randomized (1:1), controlled trial of Impella for active left ventricular unloading on top of veno-arterial extracorporeal membrane oxygenation vs. veno-arterial extracorporeal membrane oxygenation alone for the treatment of cardiogenic shock.

DETAILED DESCRIPTION:
In the past years extensive efforts in developing treatment strategies for patients with cardiogenic shock have been performed. One promising such strategy is active unloading of the left ventricle while simultaneously supporting the circulatory system with veno-arterial extracorporeal membrane oxygenation. Recently, in a multinational, multicenter, retrospective registry, it has been shown that this approach might be associated with lower mortality .

The investigators now seek to extend the evidence on this topic and to test this approach in a prospective, randomized, controlled, multicenter trial. A power calculation has been conducted based on the data from the registry. N=198 patients with cardiogenic shock will be randomized 1:1 to be either treated with an Impella for active left ventricular unloading on top of veno-arterial extracorporeal membrane oxygenation or with veno-arterial extracorporeal membrane oxygenation alone. A blinded interim analysis will be performed, which might lead to an adjustment of the enrollment target. The primary endpoint of this study will be death from any cause 30 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

Severe cardiogenic shock due to severe left ventricular dysfunction:

* Systolic blood pressure <90 mmHg or need for catecholamines to maintain such blood pressure
* Signs of impaired organ perfusion with at least one of the following: altered mental status OR cold, clammy skin OR oliguria with urine output <30 ml/h
* Arterial lactate >5 mmol/l

Exclusion Criteria:

* Post-cardiotomy cardiogenic shock.
* Cardiogenic shock due to acute rejection in heart transplant recipients.
* Obstructive cardiogenic shock (e.g. cardiogenic shock due to fulminant pulmonary embolism)
* Cardiogenic shock due to other causes (e.g. bleeding, hypothermia)
* Pre-existing Impella treatment.
* Onset of shock >12 hours.
* Mechanical complication of acute myocardial infarction.
* Prolonged resuscitation (>60 minutes).
* Severe peripheral artery disease with infeasibility for Impella or veno-arterial extracorporeal membrane oxygenation implantation.
* Age <18 or >80 years.
* Other severe concomitant disease with life expectancy <6 months.
* Participation in another trial with an intervention or pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to death from any-cause within 30 days after randomization | 30 days
  Time to death from any-cause within 30 days after randomization

SECONDARY OUTCOMES:
Death from any-cause at 6 and 12 months as well as time to death at these time points | 6 and 12 months
  Cardiovascular death at day 30, 6 months and 12 months as well as time to death at these time points
Cardiovascular death at day 30, 6 months and 12 months as well as time to death at these time points | 30 days, 6 and 12 months
  Cardiovascular death at day 30, 6 months and 12 months as well as time to death at these time points
Length of veno-arterial extracorporeal membrane oxygenation therapy, mechanical ventilation, inotrope therapy and stay at the intensive care unit (in days). | 12 months
  Length of veno-arterial extracorporeal membrane oxygenation therapy, mechanical ventilation, inotrope therapy and stay at the intensive care unit (in days).
Days free from veno-arterial extracorporeal membrane oxygenation therapy in 30 days | 30 days
  Days free from veno-arterial extracorporeal membrane oxygenation therapy in 30 days
Need for renal replacement therapy until day 30, 6 months and 12 months | 30 days, 6 and 12 months
  Need for renal replacement therapy, intermittent or ongoing, until day 30, 6 months and 12 months
Neurological function (per Cerebral Performance Category) at day 30, 6 months and 12 months | 30 days, 6 and 12 months
  Neurological function (per Cerebral Performance Category) at day 30, 6 months and 12 months
Rate of incidence of hospitalization for heart failure (hospitalization for more than 24 hours with heart failure as the main reason) as well as time to first event after 6 months and 12 months and recurrent events within 12 months | 6 and 12 months
  Rate of incidence of hospitalization for heart failure (hospitalization for more than 24 hours with heart failure as the main reason) as well as time to first event after 6 months and 12 months and recurrent events within 12 months
Left ventricular function assessed by echocardiography at day 30, 6 months and 12 months | 30 days, 6 and 12 months
  Left ventricular function assessed by echocardiography at day 30, 6 months and 12 months
Quality of life as assessed by the "Kansas City Cardiomyopathy Questionnaire" at 30-days and at 12 months | 30 days and 6 months
  Quality of life as assessed by the "Kansas City Cardiomyopathy Questionnaire" at 30-days and at 12 months
6-Minute Walking Distance at day 30, 6 months and 12 months | 30 days, 6 and 12 months
  6-Minute Walking Distance at day 30, 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Heart and Vascular Center Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moussa MD, Roux J, Jungling M, Ramdane N, Loobuyck V, Brassart B, Rousse N, Dupre C, Mugnier A, Khalipha A, Bardeesi ASA, Lukowiak O, Lefebvre L, Juthier F, Robin E, Labreuche J, Thellier L, Vincentelli A. Impella Versus Selective Biatrial Canulation for Left Ventricular Unloading During Extracorporeal Membrane Oxygenation. Cardiovasc Ther. 2026 Feb 8;2026:3669575. doi: 10.1155/cdr/3669575. eCollection 2026. PMID 41668891
- [Derived] Schrage B, Sundermeyer J, Blankenberg S, Colson P, Eckner D, Eden M, Eitel I, Frank D, Frey N, Graf T, Kirchhof P, Kupka D, Landmesser U, Linke A, Majunke N, Mangner N, Maniuc O, Mierke J, Mobius-Winkler S, Morrow DA, Mourad M, Nordbeck P, Orban M, Pappalardo F, Patel SM, Pauschinger M, Pazzanese V, Radakovic D, Schulze PC, Scherer C, Schwinger RHG, Skurk C, Thiele H, Varshney A, Wechsler L, Westermann D. Timing of Active Left Ventricular Unloading in Patients on Venoarterial Extracorporeal Membrane Oxygenation Therapy. JACC Heart Fail. 2023 Mar;11(3):321-330. doi: 10.1016/j.jchf.2022.11.005. Epub 2023 Jan 11. PMID 36724180